CLINICAL TRIAL: NCT04902261
Title: Prospective Exploratory Study of Tislelizumab Combined With Nab-paclitaxel and Gemcitabine for Postoperative Recurrence of Pancreatic Cancer
Brief Title: Tislelizumab Combined With Nab-paclitaxel and Gemcitabine for Recurrent Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Guo ShiWei, Principal Investigator, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2020-144
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Recurrent Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tislelizumab; Taxes; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab combined with Nab-paclitaxel and Gemcitabine (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Nab paclitaxel; Drug: Gemcitabine
- Nab-paclitaxel and Gemcitabine (Active Comparator)
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200 mg every three weeks
  Arms: Tislelizumab combined with Nab-paclitaxel and Gemcitabine
Drug: Nab paclitaxel — Nab-paclitaxel 125mg/m2 on d1 and d8 every three weeks
Drug: Gemcitabine — Gemcitabine 1000mg/m2 on d1 and d8 every three weeks

SUMMARY:
To evaluate the efficacy of Tislelizumab combined with Nab-paclitaxel and Gemcitabine in the treatment of recurrent pancreatic cancer

DETAILED DESCRIPTION:
There is heterogeneity in desmoplasia between different metastatic sites in pancreatic cancer. The tumor quasi-characteristics of patients with metastatic PDAC at presentation were more obvious than those of epithelial characteristics, and the quasi-and epithelial subtypes showed different responses to chemotherapy regimens, and the epithelial phenotype tumor quasi-phenotype was associated with metastasis-free survival. Therefore, different metastases of pancreatic cancer may respond differently to medical treatment. There were different metastases after postoperative recurrence of pancreatic cancer, 25.2% had only liver metastases, 14.7% had only lung metastases, 14.7% had multiple distant metastases, and about more than half of the patients had postoperative recurrence with only distant metastases and no in situ metastasis. Then whether there is a difference in the efficacy of PD1 drug therapy in patients with different metastases needs to be further verified.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiologically or histologically confirmed postoperative Recurrent Pancreatic Cancer
* Patients with at least one measurable lesion (according to RECIST 1.1 criteria);
* Have not received gemcitabine-based regimen after surgery
* No systemic treatment after diagnosis of recurrence
* ECOG score 0-1
* Expected survival ≥ 3 months;
* Liver function is essentially normal: absolute neutrophil count > 1500/mm ³; platelet count > 100,000/mm ³; creatinine less than 1.5 times the upper limit of normal or calculated creatinine clearance (CRCI) > 45 mL/min; total bilirubin ≤ 2.0 mg/dL; aspartate aminotransferase (AST) and alanine aminotransferase less than 2.5 times the upper limit of normal
* Appropriate to participate in this trial as assessed by the investigator before entering the study
* Male and female subjects of childbearing potential must agree to use an effective method of contraception throughout the study
* Signed Informed Consent Form

Exclusion Criteria:

* Patients who only undergo abdominal laparotomy but do not undergo resection of pancreatic tumor tissue
* Received gemcitabine-based regimen after surgery
* Systemic treatment after diagnosis of recurrence
* Patients with previous allergic reactions to similar drugs
* Pregnant or lactating patients
* Presence of pericardial effusion, uncontrolled pleural effusion, or clinically significant ascites at screening (including detectable ascites or ascites requiring puncture and aspiration on physical examination at screening)
* History of interstitial lung disease, pneumonitis, or uncontrolled systemic disease, including diabetes, hypertension, pulmonary fibrosis, acute lung disease, etc
* Patients with severe cardiovascular diseases within 12 months before enrollment, such as symptomatic coronary heart disease, ≥ grade II congestive heart failure, uncontrolled arrhythmia, myocardial infarction, etc
* Presence of any active immunodeficiency or autoimmune disease and/or history of any immunodeficiency or autoimmune disease that may recur at screening (e.g., hypothyroidism or hyperthyroidism, interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, etc)
* Use of steroids or other systemic immunosuppressive therapy 14 days prior to enrollment
* Patients with other previous malignancies who are not cured
* Immunodeficient patients, such as HIV-positive
* Uncontrollable psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-11-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
1-Year Survival Rates | Up to 2 years
  The proportion of patients who survive more than 1 year after treatment.

SECONDARY OUTCOMES:
Overall Response Rate（ORR) | Up to 2 years
  the proportion of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR)
Progression Free Survival (PFS) | Up to 2 years
  The time from the date of treatment to the first of either disease progression, relapse or death
Overall survival (OS) | Up to 2 years
  The time from the date of treatment start to the date of death or to the date of last follow-up for patients alive
Adverse Events (AEs) | Up to 2 years
  the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0; Surgical safety including Intraoperative blood loss，PHLF assessed by ISGLS（2012），Postoperative complications evaluated by modified Clavien-Dindo system.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Jin, Doctor, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No